CLINICAL TRIAL: NCT07187388
Title: The Impact of Transcutaneous Electrical Stimulation on Facial Pain, Jaw Mobility, and Oral Health in Individuals With Motor Neuron Disease.
Brief Title: Investigating the Impact of Electrical Stimulation on Facial Pain, Jaw Movement and Oral Health in People With Motor Neuron Disease.
Acronym: MND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-356-NSU
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Primary Lateral Sclerosis (PLS); Motor Neuron Disease, Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; ALS; PLS; Motor Neuron Disease; MND; Facial Pain; jaw pain
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Facial Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transcutaneous electrical stimulation to reduce facial pain and improve jaw ROM in ALS and PLS. (Experimental): All 10 participants will receive a single TENS intervention, with electrodes placed over the masseter and TMJ regions. This intervention is designed to evaluate TENS as a potential treatment for reducing facial pain and improving jaw mobility and chewing function in individuals with ALS and PLS..
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation to reduce facial pain and improve jaw range of motion in ALS and PLS

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation to reduce facial pain and improve jaw range of motion in ALS and PLS — TENS intervention will be administered using a current-controlled TENS device that produces charge-balanced, symmetrical biphasic rectangular pulses. Participants will be seated and skin cleaned prior to applying 2 self-adhesive round surface electrodes (25mm) on each side of the face. One electrode (anode) will be placed over the masseter muscle belly, while the other (cathode) will be positioned over the TMJ. Electrode placement will be confirmed by palpation of the TMJ and Masseter. This set up will be mirrored on the opposite side. Once all 4 electrodes are in place, the TENS unit will be turned on.
  Participants will remain seated. The TENS unit will be set to manual mode to deliver the stimulation at a frequency of 50 Hertz (Hz) and a pulse width of 200 microseconds (µseconds). Stimulation amplitudes will be gradually increased from 0 milliamps (mA) to each participant's tolerance level. The 30 minute TENS intervention will then take place.

SUMMARY:
The goal of this clinical trial is to evaluate the impact of non-invasive electrical stimulation, when placed on the facial muscles can reduce facial pain and improve jaw mobility, and chewing in individuals with Amyotrophic Lateral Sclerosis (ALS) and Primary Lateral Sclerosis (PLS). The secondary goal is to evaluate the impact of non-invasive electrical stimulation on patient reported difficulty performing oral hygiene tasks in individuals with ALS and PLS. Participants will attend one in-person clinic visit and participate in one telephone interview 24 hours after the treatment. The clinic visit will include pre-intervention assessments, a single 30-minute treatment of electrical stimulation followed by post-intervention assessments.

The assessments will include a self-rating of jaw and facial pain, a range of motion test where participants will be asked to open their jaw as wide and as far to the side as possible, and a chewing efficiency test using a saltine cracker. Twenty-four hours later, participants will receive a follow-up phone call to self-rate their facial pain and report any difficulty performing oral hygiene tasks.

The treatment consists of a single 30-minute electrical stimulation session. Electrode pads will be placed on the participant's facial region, specifically over the masseter muscle belly and the TMJ area, while the participant is seated comfortably. The pads will be connected to an FDA-approved electrical stimulator, and the current will be adjusted to the participant's comfort level. Once set, the participant will remain seated for 30 minutes. At the end of the session, the stimulator will be turned off and the electrode pads removed.

DETAILED DESCRIPTION:
In this prospective, cross-sectional study, individuals with ALS and PLS will participate in one in-person clinic visit, followed by a telephone interview 24 hours post-treatment. During the clinic visit, pre-intervention assessments will be conducted to evaluate facial pain, jaw range of motion (jROM), mastication efficiency, and patient-reported difficulty with oral hygiene tasks. Following these assessments, participants will receive a single 30-minute TENS treatment. The PI or Co-PI will be present throughout the intervention, monitoring for any discomfort and providing participants the option to discontinue treatment if needed using a predetermined signal.

Post-intervention assessments, identical to the pre-intervention evaluations, will then take place. The entire clinic visit is expected to take approximately 90 minutes. A brief telephone interview 24 hours after the intervention will collect subjective feedback, including patient-reported pain levels and perceived difficulty of performing oral hygiene tasks.

The primary outcome measure will be patient-reported pain, defined by the International Association for the Study of Pain "an unpleasant sensory and emotional experience associated with, or resembling that associated with, actual or potential tissue damage," localized to the jaw region and assessed using a Numeric Rating Scale (NRS). Secondary outcome measures will include jROM, the ability to chew solid foods, and participants' perceived difficulty with oral hygiene tasks, as outlined below.

Participants.

Participants will be identified and recruited during weekly ALS/PLS multidisciplinary clinic visits. The study will enroll 10 pALS/pPLS between the ages of 25 and 90.

METHODS Pre-Intervention Assessment: Estimated Time 25 minutes

1. Jaw Pain Assessment:

   Pain levels will be assessed using the NRS scale. This scale uses a 0-10 numeric range, where 0 represents no pain and 10 represents the worst possible pain. Participants will rate their pain by choosing a number between 0 and 10 to indicate their pain intensity pre-, post-, and 24 hours post-intervention.
2. Jaw Range of Motion Assessment To measure maximal incisal opening (oral opening), the TheraBite range of motion (ROM) scale will be used. The TheraBite ROM scale is a disposable tool that assists investigators to assess the distance in millimeters (mm) between the upper and lower central incisors when the patient opens their mouth as wide as possible or performs lateral jaw movements. Maximum interincisal distance (MID) and Maximal lateral jaw movement will be measured in mm both pre- and post- intervention.

   The participant will be instructed to open their mouth as wide as possible within a pain-free range. The TheraBite ROM Scale will be positioned between the upper and lower central incisors, and the maximum opening will be measured in millimeters (mm).

   The participant will be instructed to move their jaw sideways to the left and right within a pain-free range. The TheraBite ROM Scale will be used to measure the distance between the midline of the upper and lower teeth, with the values recorded in millimeters (mm).

   A surface EMG sensor will be positioned on the masseter muscle belly during both jROM assessments to measure muscle activity at rest, during passive stretch and during muscle activation. This will provide real-time data visualization to quantify muscle activation patterns pre- and post- intervention.
3. Mastication Efficiency Assessment : Test of Mastication and Swallowing Solids (TOMASS)

The TOMASS will be utilized to assess solid bolus ingestion by quantifying masticatory efficiency, speed, and safety, providing objective measurements of mastication performance. The objective outcomes include the number of masticatory cycles and swallows per bite, and duration.

3b. Oral Transit Time (OTT)

In the event the participant cannot chew a saltine cracker, required for the TOMASS, the OTT will be utilized. The OTT is a tool to quantify how many seconds it takes a participant to consume a modified textured food item (IDDSI level 4, apple sauce) and clear bolus from oral cavity. OTT will be described using quantitative parameters from the Mann Assessment of Swallowing Ability (MASA): Score of 2 = No oral transit movement observed; Score of 4 = delay >10 seconds ; Score of 6 =delay > 5 seconds; Score of 8 = delay >1 second; Score of 10 = no OTT delay.

4. Oral Hygiene - Numerical Rating Scale (NRS)

Patient-reported difficulty completing oral hygiene will be assessed using a NRS ranging from 0 (no difficulty) to 10 (significant difficulty). Participants will rate their perceived difficulty pre-intervention and 24 hours post intervention.

5. TENS Intervention - 40 minutes

TENS intervention will be administered using a current-controlled TENS device that produces charge-balanced, symmetrical biphasic rectangular pulses. Participants will be seated and skin cleaned prior to applying 2 self-adhesive round surface electrodes (25mm) on each side of the face. One electrode (anode) will be placed over the masseter muscle belly, while the other (cathode) will be positioned over the TMJ. Electrode placement will be confirmed by palpation of the TMJ and Masseter. This set up will be mirrored on the opposite side. Once all 4 electrodes are in place, the TENS unit will be turned on. This is estimated to take 10 minutes.

Participants will remain seated. The TENS unit will be set to manual mode to deliver the stimulation at a frequency of 50 Hertz (Hz) and a pulse width of 200 microseconds (µseconds). Stimulation amplitudes will be gradually increased from 0 milliamps (mA) to each participant's tolerance level. Participants will be instructed to indicate when the stimulation feels "strong but comfortable." The tolerated mA level will be recorded and maintained for the full 30-minute session.

The PI or Co-PI will be present throughout the intervention, monitoring for any discomfort and providing participants the option to discontinue treatment if needed. At the end of the session, the TENS device will be powered off, electrodes will be removed, and post-intervention testing will be conducted.

6. Post Intervention Assessments are identical to pre-intervention assessments and are estimated to take 25 minutes.

7. 24 hour telephone interview - Estimated time - 10 minutes. The participant will be contacted 24 hours after completion of intervention and a telephone interview will be conducted. The PI or co-PI will contact the participant and collect subjective feedback, including patient reported pain levels, perceived difficulty of performing oral hygiene tasks, both rated utilizing the NRS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, probable, or definite ALS (El-Escorial Revisited) OR diagnosis of definite PLS by the treating neurologist and based on the consensus diagnostic criteria for PLS
* Subjective report of jaw pain, indicated by a NRS score of > or = 3/10.

Exclusion Criteria:

* history of head or neck cancer
* history of CVA
* history of past facial surgery with hardware placement
* history of pacemaker
* diagnosis of significant cognitive impairment by the treating physician
* history of seizures or diagnosis of epilepsy
* open wound at the area of electrode placement
* complete loss of sensation at the area of electrode placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-08-13 (Estimated); Study Completion 2026-08-13 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale for Pain | Baseline, immediately post-intervention and 24 hours post-intervention
  0-10 numeric rating scale where participants will self rate their pain on a scale of 0-10 with 0 = no pain and 10 = worst possible pain.

SECONDARY OUTCOMES:
Jaw Range of Motion (jROM) Assessment | Baseline and immediately post-intervention
  Maximum interincisal distance (MID) and Maximal lateral jaw movement will be measured utilizing the TheraBite range of motion scale. The participant will be instructed to open their mouth as wide as possible within a pain-free range. The TheraBite ROM Scale will be positioned between the upper and lower central incisors, and the maximum opening will be measured in millimeters (mm). The participant will be instructed to move their jaw sideways to the left and right within a pain-free range. The TheraBite ROM Scale will be used to measure the distance between the midline of the upper and lower teeth, with the values recorded in millimeters (mm). A surface EMG sensor will be positioned on the masseter muscle belly during both jROM assessments to measure muscle activity at rest, during passive stretch and during muscle activation. This will provide real-time data visualization to quantify muscle activation patterns pre- and post- intervention.
Test of Mastication and Swallowing Solids (TOMASS) | Baseline and immediately post-intervention
  The TOMASS will be utilized to assess solid bolus ingestion by quantifying masticatory efficiency, speed, and safety, providing objective measurements of mastication performance. The TOMASS allows clinicians to capture detailed information about the relationship between jaw function, pain, and mastication issues when consuming a standardized solid food item (saltine cracker). The objective outcomes include the number of masticatory cycles and swallows per bite, and duration.
Numeric Rating Scale for Oral Hygiene | Baseline and 24 hours post intervention.
  Patient-reported difficulty completing oral hygiene will be assessed using a NRS ranging from 0 (no difficulty) to 10 (significant difficulty). Participants will rate their perceived difficulty by providing a number from 0 (no difficulty) to 10 (significant difficulty).

OTHER OUTCOMES:
Oral Transit Time (OTT) | Baseline and immediately post-intervention
  In the event the participant cannot chew a saltine cracker, required for the TOMASS, the OTT will be utilized. The OTT is a tool to quantify how many seconds it takes a participant to consume a modified textured food item (IDDSI level 4, apple sauce) and clear bolus from oral cavity. OTT will be described using quantitative parameters from the Mann Assessment of Swallowing Ability (MASA): Score of 2 = No oral transit movement observed; Score of 4 = delay >10 seconds ; Score of 6 =delay > 5 seconds; Score of 8 = delay >1 second; Score of 10 = no OTT delay.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Southeastern University, David and Cathy Husman Neuroscience Institute, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All 10 participants baseline assessments, post assessments and 24 hour interview responses will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD will be available 12 months after publication of the primary results and for a period of 5 years.
Access Criteria: De-identified IPD will be shared with qualified researchers upon reasonable request, subject to review by the study investigators and execution of a data use agreement.

REFERENCES:
- [Background] Alizadeh A, Karagah A, Tabrizi R, Shadman L, Arjmand A, Tofangchiha M, Patini R. Effect of transcutaneous electrical nerve stimulation on pain, edema, and trismus after surgical removal of impacted third molars: a split-mouth randomized clinical trial. Med Oral Patol Oral Cir Bucal. 2024 Mar 1;29(2):e211-e218. doi: 10.4317/medoral.26193. PMID 37823292
- [Background] Zayan K, Felix ER, Galor A. Transcutaneous Electrical Nerve Stimulation for Facial Pain. Prog Neurol Surg. 2020;35:35-44. doi: 10.1159/000509620. Epub 2020 Jul 21. PMID 32694253
- [Background] Shanavas M, Chatra L, Shenai P, Rao PK, Jagathish V, Kumar SP, Naduvakkattu B. Transcutaneous electrical nerve stimulation therapy: An adjuvant pain controlling modality in TMD patients - A clinical study. Dent Res J (Isfahan). 2014 Nov;11(6):676-9. PMID 25540662
- See also: Link to TENS device utilized — https://www.tenspros.com/intensity-select-combo-ii-tens-ems-if-russian-stim-di2195.html?srsltid=AfmBOop7EXKQ0zq6G2FVWZDkZzaZriGKL9YatZStCTIc2CiSxvuWXuNt
- See also: EMG surface sensor — https://quickstart.k-invent.com/wp-content/uploads/2024/11/K-MYO-manual-V3_ENG_2024-10-11web.pdf